CLINICAL TRIAL: NCT07162337
Title: BILMOD: BILe Acid-gut Microbiome Axis MODification Through Diet Education for Colorectal Cancer Prevention
Brief Title: BILe Acid-gut Microbiome Axis MODification Through Diet Education for Colorectal Cancer Prevention
Acronym: BILMOD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew T. Chan, MD, MPH, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-611
Record Dates: First submitted 2025-07-31; First posted 2025-09-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer Prevention; Colorectal Adenoma
Keywords: colorectal cancer; colorectal cancer prevention; colorectal adenoma; obesity; western diet
MeSH Terms: conditions — Colorectal Neoplasms; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Increased Plant-Based Diet and Decreased Animal-Based Diet (Experimental): Participants will be instructed to self-regulate their diet by increasing the amount of plant-based foods while decreasing the amount of animal-based foods for a 4-week period.
  Interventions: Behavioral: Increased Plant-Based Diet and Decreased Animal-Based Diet

INTERVENTIONS:
Behavioral: Increased Plant-Based Diet and Decreased Animal-Based Diet — Self-regulated diet; increased plant-based foods with decreased animal-based foods

SUMMARY:
This research study is a prospective, single-arm clinical trial to assess the effect of a dietary intervention for more plant-based and less animal-based food intake on secondary bile acid production, gut microbiota, circulating biomarkers and gene expression associated with colonic bile acid receptor activation and colorectal cancer.

DETAILED DESCRIPTION:
In this research study, the investigators are:

* Investigating the effect of more plant-based and less animal-based food intake on bile acid metabolomic composition in stool among individuals with a history of colorectal adenoma.
* Investigating the effect of more plant-based and less animal-based food intake on plasma bile acid metabolomic composition, the gut microbiome, circulating biomarkers and gene expression associated with colonic bile acid receptor activation and colorectal cancer among individuals with a history of colorectal adenoma.

Based on the following evidence:

* Growing evidence indicates that the gut microbiome and its metabolites play important roles in mediating the dietary effects on colorectal cancer risk
* Secondary bile acids are increasingly appreciated as important metabolites underlying the metabolic link between Western diet, the gut microbiome, and colorectal cancer
* Evidence suggests that secondary bile acids trigger a plethora of tumorigenic effects in the colon, including inflammation, oxidative DNA damage, and apoptosis resistance
* Epidemiological studies have revealed that a higher circulating level of secondary bile acids, particularly deoxycholic acid and lithocholic acid, was associated with an increased risk of colorectal cancer
* High fat intake has been repeatedly reported to increase secondary bile acids, but the findings on how other nutrients or foods in Western diet may influence secondary bile acids remain mixed

The research procedures include screening for eligibility, study intervention, and scheduling two clinical research visits:

* Initial visit - immediately before starting the dietary intervention
* 1 week of observation prior to dietary intervention
* 4 weeks of dietary intervention (increasing plant based food and reducing animal-based food)
* Final visit (after completing the dietary intervention)

At the Initial and Final visits, there will be a collection of lifestyle and nutritional questionnaire data, blood samples, and stool samples. The initial visit will establish the baseline data. The 1-week pre-intervention observation will establish baseline food diary data (every 2 days). The 4-week intervention phase will involve phone calls from study staff to guide participants in their diet changes, additional food diary entries (every 2 days), stool sample collection (every 7 days), and body weight reporting (every 7 days).

It is expected that about 40 people will take part in this research study.

This research is being supported by the National Cancer Institute.

ELIGIBILITY:
Inclusion Criteria:

* Underwent screening or surveillance colonoscopy with removal of at least one adenoma.
* Age 18-80 years.
* Habitually consume a Western pattern diet.
* BMI of at least 18.5 kg/m2 but less than 35 kg/m2
* Weight stable in last 3 months (loss or gain <4%).
* Subjects must be able and willing to follow study procedures and instructions.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Strict dietary patterns (e.g., vegan, carnivore, kosher, low-carb etc.).
* Diagnosis of inflammatory bowel disease, liver or kidney disease, bleeding diathesis.
* Any prior diagnosis of gastrointestinal cancer (including esophageal, small intestine, colon, pancreatic), or any diagnosis of other cancers (with the exception of nonmelanoma skin) in which there has been any active treatment within the last three years.
* Known diagnosis of Familial Adenomatous Polyposis (FAP) or Hereditary Non-Polyposis Colorectal Cancer (HNPCC, Lynch Syndrome).
* Any adenoma that was not completely removed during previous colonoscopy.
* Known bleeding tendency/condition (e.g. von Willebrand disease) or history of peptic ulcer or gastrointestinal bleed requiring hospitalization, endoscopic complications, or contraindication to colonoscopy.
* Current use of anticoagulant therapies, including Heparin, Warfarin, Dalteparin sodium, Bivalirudin, Argatroban, Lepirudin, Heparin Sodium, Heparin/Dextrose, and an unwillingness or inability to discontinue anticoagulants.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Regular use of aspirin.
* Use of antibiotics or probiotics.
* Inability or unwillingness to abstain from limited consumption of animal-based food or to provide blood or stool samples during the study.
* Participants who are receiving any other investigational agents.
* Pregnant or breastfeeding.
* Known positive test for human immunodeficiency virus (HIV), hepatitis C virus, or acute or chronic hepatitis B infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Stool Metabolomics | From Baseline to Final Visit (5 weeks)
  Comparing change in stool metabolomics, using non-targeted global metabolomics analysis on stool samples to examine intensity changes in the stool metabolite profile.

SECONDARY OUTCOMES:
Relative Composition of Gut Microbiome | From Baseline to Final Visit (5 weeks)
  Comparing change in gut microbiome features (species - to strain level specificity; metabolic pathways; enzymes) and metabolites using deep meta'omic profiling in pre- and post- treatment samples.

OTHER OUTCOMES:
Change in Plasma Bile Acid Metabolomics | From Baseline to Final Visit (5 weeks)
  Comparing change in plasma bile acid metabolomics, using non-targeted global metabolomics analysis on stool samples to examine intensity changes in the stool metabolite profile.
Relative Composition of Circulating Biomarkers | From Baseline to Final Visit (5 weeks)
  The investigators will use plasma collected in EDTA tubes and processed within 2-4 hours of collection to measure circulating protein biomarkers associated with bile acid receptor activity, including plasma concentrations of 92 inflammation-related proteins measured using the proximity extension immunoassay [PEA] technology [Olink Proteomics®, Uppsala, Sweden] with the ProSeek Multiplex Inflammation panel (Olink® target 92 inflammation panel). These measurements will be performed on samples collected at the initial and final visits to evaluate diet-induced changes in bile acid signaling.
Relative Composition of Circulating Gene Expression Profile | From Baseline to Final Visit (5 weeks)
  The investigators will use plasma collected in EDTA tubes and processed within 2-4 hours of collection to measure circulating biomarkers associated with colorectal tumorigenesis using validated enzyme-linked immunosorbent assay (ELISA) kits, including BIRC5 (survivin), FOXM1, MYC, IL6, TNF, and S100A8/A9. These measurements will be performed on samples collected at the initial and final visits to evaluate diet-induced changes in systemic inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T. Chan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Andrew T. Chan, MD, MPH. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the MGB Innovation at PHSINNOVATIONSUPPORT@partners.org